CLINICAL TRIAL: NCT04772573
Title: The Treatment Challenges and Limitation in High-Voltage Pediatric Electrical Burn at Rural Area: A Case Report
Brief Title: The Treatment Challenges and Limitation in High-Voltage Pediatric Electrical Burn at Rural Area
Status: Completed | Type: Observational
Sponsor: S.K. Lerik General Hospital (Other)
Responsible Party: Principal Investigator, Kevin Leonard Suryadinata, MD, S.K. Lerik General Hospital
Other Study IDs: SKL002
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Burns; Electrical Burn; Burn Degree Second; Burn Scar
MeSH Terms: conditions — Burns; Burns, Electric

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A case of high-voltage pediatric electrical burn involving a fully conscious 13-year old boy who was admitted to the emergency room after being electrocuted by high-voltage power cable, with superficial partial thickness burn over right arm, trunk, and left leg (26% of total body surface area) with cardiac abnormality e.g. tachycardia and non-specific ST depression. Treatments were based on Australian New Zealand Burns Association algorithm with several modifications, i.e. administering lower concentration of oxygen with nasal cannula instead of non-rebreathing mask and intravenous Ketorolac and Metamizole as analgesic instead of morphine due to limitation in infrastructure and knowledge. The patient underwent surgical debridement and strict observation with no signs of abnormality found during hospital stay. Wound dressing consisted of silver sulfadiazine, Sofra-tulle® and dry sterile gauze were used until epithelialization. After the wound healed, the patient resumed wearing elastic bandage and moisturizer on the wound area. The patient was observed daily through 7 days of hospitalization and followed-up for 1 year, achieving normal physiologic function of the affected area but unsatisfactory esthetic result. This case report showed that there is still a lack of burn prevention programs in the rural area, resulted in inadequate first aid application for electrical burn. There is a need for acknowledging and maximizing the implementation of available standardized guidelines e.g. Australian New Zealand Burns Association by giving homogenized training to personnel as well as providing feasible equipment, and then followed by strict monitoring for the patient. The focus of the burn program should also include burn rehabilitation, psychosocial needs and any complaints needing expert opinion in an outpatient setting in addition to adequate burn management for life saving and good wound healing.

ELIGIBILITY:
Inclusion Criteria:

* patient with acute electrical burn wound

Exclusion Criteria:

* patient does not want to participate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with acute electrical burn wound
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Wound healing | 1 month
  The healing rate of burn wound

SECONDARY OUTCOMES:
Burn Scar | 1 year
  The appearance and function of the scar and the affected areas

CONTACTS AND LOCATIONS:
Overall Officials: Adi Basuki, MD, Principal Investigator — S.K.Lerik Public Hospital
Locations (1):
- S.K.Lerik General Hospital, Kupang, East Nusa Tenggara, Indonesia